CLINICAL TRIAL: NCT04864548
Title: A Dose Finding Human Experimental Infection Study With SARS-CoV-2 in Healthy Volunteers With Immunologically Sensitised With Either Previous, SARS-CoV-2 Infection and/or Vaccination Against SARS-CoV2
Brief Title: COV-CHIM01: SARS-CoV-2 (COVID-19) Dose Finding Infection Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: COV-CHIM01
Record Dates: First submitted 2021-04-20; First posted 2021-04-29 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus
Keywords: Covid-19; SARS-CoV-2; Controlled human infection model; Infection study
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Masking Description: This is an open-label trial, however in order to minimise volunteer adverse event reporting bias by volunteers, study participants will be kept blinded to swab results for as long as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Group 1A: Low dose challenge (Experimental): Intranasal viral challenge with 1 x 10^1 TCID_50 in previously infected volunteers
  N= 6-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 1B: Medium dose #1 challenge (Experimental): Intranasal viral challenge with 1 x 10^2 TCID_50 in previously infected volunteers
  N= 6-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 1C: Medium dose #2 challenge (Experimental): Intranasal viral challenge with 1 x 10^3 TCID_50 in previously infected volunteers
  N= 6-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 1D: Medium dose #3 challenge (Experimental): Intranasal viral challenge with 1 x 10^4 TCID_50 in previously infected volunteers
  N= 4-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 1E: High dose challenge (Experimental): Intranasal viral challenge with 1 x 10^5 TCID_50 in previously infected volunteers
  N= 4-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 2: Safety & Dose confirmation Group (Experimental): Intranasal viral challenge with the dose identified from Group 1a-e (1x10^1, 1x10^2, 1x10^3, 1x10^4, or 1x10^5 TCID_50)
  N=10-30 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 3a: Medium dose #1 challenge (Experimental): Intranasal viral challenge with 1 x 10^2 TCID_50 in previously uninfected, vaccinated volunteers
  N=6-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 3b: Medium dose #2 challenge (Experimental): Intranasal viral challenge with 1 x 10^3 TCID_50 in previously uninfected, vaccinated volunteers
  N=4-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 3c: Medium dose #3 challenge (Experimental): Intranasal viral challenge with 1 x 10^4 TCID_50 in previously uninfected, vaccinated volunteers
  N=4-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 3d: High dose challenge (Experimental): Intranasal viral challenge with 1 x 10^5 TCID_50 in previously uninfected, vaccinated volunteers
  N=4-8 participants
  Interventions: Biological: SARS-CoV-2 virus
- Group 4: Safety & Dose confirmation Group (Experimental): Intranasal viral challenge with the dose identified from Group 3a-d (1x10^2, 1x10^3, 1x10^4 or 1x10^5 TCID_50)
  N=10-30 participants
  Interventions: Biological: SARS-CoV-2 virus

INTERVENTIONS:
Biological: SARS-CoV-2 virus — The SARS-COV-2 challenge virus strain was originally obtained from a nose/throat swab taken from a patient who developed respiratory symptoms consistent with COVID-19. The isolate was plaque purified to obtain a 'single' virus entity. The selected plaque, B1, was subsequently manufactured in accordance with GMP at the Great Ormond Street manufacturing suite.

SUMMARY:
A phase I, experimental dose finding, open label, clinical infection, safety and viral detection optimisation in previously SARS-CoV-2 infected (unvaccinated or vaccinated) or uninfected vaccinated volunteers.

DETAILED DESCRIPTION:
This is a phase I dose escalation challenge study in which increasing titres of wild-type SARS-CoV-2 (1x10^1 TCID_50, 1x10^2TCID_50, 1x10^3TCID_50, 1x10^4TCID_50 and 1x10^5TCID_50) will be administered intranasally to different groups of volunteers in order to achieve a 50% (+/-10%) attack rate as determined by quantitative live viral detection and/or qPCR detection in naso-pharyngeal secretions at two consecutive 12 hourly time points (at least 24 hours after inoculation). Dose escalation will be capped at 10^5 TCID50 and we will proceed to dose confirmation, following DSMB safety review, even if we do not meet our target attack rate of 50% +/- 10%, to enable a larger sample size to assess the dynamic range of protection at that dose and ensure confidence in the negative infection rate at that dose.

A Data Safety Monitoring Board (DSMB) will review safety and quantitative virology at each dose level and will recommend continuation based on emergent data.

Rescue treatment with a single course of oral Paxlovid will commence immediately after any warning symptoms or signs of COVID-19 disease beyond mild disease.

Once the optimal dose of wildtype SARS-CoV-2 has been identified for previously infected volunteers and uninfected vaccinated volunteers (dose escalation groups 1 and 3), further challenge infections in groups 2 and 4 may proceed.

Volunteers will remain in isolation rooms within the clinical trials unit for a minimum of 14 days post inoculation and until demonstration of the absence of live virus in two sequential samples. All 4 groups will together enrol up to 132 volunteers.

This study will be funded by the Wellcome Trust and Department of Health and Social Care (DHSC).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-30 years on proposed date of enrolment.
2. Body Mass Index (BMI) ≥18.5 kg/m2and ≤28 kg/m2.
3. In good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with subject safety, as defined by medical history, physical examination, routine laboratory tests, cardiovascular magnetic resonance imaging or echocardiogram, ECG, pulmonary function tests and Chest X-Ray as determined by the Investigator at a screening evaluation.
4. Volunteer is willing and able to give written informed consent for participation in the study
5. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner or any relevant health authority
6. Allow the investigator to register volunteer details with a confidential database (The Over-volunteering Prevention Service) to prevent concurrent entry into clinical studies/trials
7. Agreement to refrain from blood donation during the course of the study
8. a. For women of child bearing potential (WOCBP), a willingness to practice continuous effective contraception during the study and, a negative pregnancy test on the day(s) of screening and challenge b. b. For women of child bearing potential (WOCBP) taking the combined oral contraceptive pill, a willingness to use barrier contraception with spermicide during treatment with Paxlovid and for 30 days after completing Paxlovid treatment (should they receive it).
9. Able and willing (in the investigator's opinion) to comply with all study requirements
10. No clinically relevant findings in medical history or on physical examination in the opinion of a clinically qualified investigator, in discussion with the CI if needed
11. For Groups 1 & 2: Previous microbiological confirmation of SARS-CoV-2 infection > 3 months prior to enrolment (Proof of positive PCR or lateral flow antigen test confirmed via medical notes/ or UK HSA or a history from a volunteer consistent with SARS-CoV-2 infection with other evidence of this infection such as a photograph of a positive lateral flow test on the volunteer's phone or similar) OR serological confirmation such as positive anti-nucleocapsid IgG serology (unless this is explainable by prior vaccination) with the most recent history of symptoms or exposure likely to represent SARS-CoV-2 infection having occurred > 3 months prior to enrolment.
12. For Groups 3 & 4: Written or electronic evidence of at least one vaccination against SARS- CoV-2 >21 days prior to enrolment (proof required would include written or electronic evidence from GP/ medical records or electronic NHS COVID pass) where no history of symptoms or exposure can be identified to determine the timing of SARS-CoV-2 infection, volunteers may be enrolled >7 weeks from the identification of anti-nucleocapsid positivity and >3 months from their last negative anti-nucleocapsid antibody test.

Exclusion Criteria:

1) History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory (excluding SARS CoV-2 infection), dermatological, gastrointestinal, endocrine, haematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological or psychiatric illness. Specifically:

1. Volunteers with any history of physician diagnosed and/or objective test confirmed asthma, chronic obstructive pulmonary disease, pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology or who have experienced:

   i) Significant/severe wheeze in the past ii) Clinically significant respiratory symptoms including wheeze which has ever resulted in hospitalisation iii) Known bronchial hyper reactivity to viruses
2. History of thromboembolic, cardiovascular or cerebrovascular disease
3. History or evidence of diabetes mellitus (Type I or Type II)
4. Any concurrent serious illness including history of malignancy that could interfere with the aims of the study or a subject completing the study. Basal cell carcinoma within 5 years of treatment or with evidence of recurrence is also an exclusion.
5. Migraine with associated neurological symptoms such as hemiplegia or vision loss. Cluster headache/migraine or prophylactic treatment for migraine
6. History or evidence of clinically significant autoimmune disease or known immunodeficiency of any cause (including HIV).
7. History of severe psychiatric illness at any time (e.g. inpatient stay, psychosis) or current significant active symptoms of anxiety and/or depression or significant claustrophobia. Consider exclusion in the following cases:

   i) Volunteers with history of anxiety related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥5 ii) Volunteers with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire-9 score is ≥4 iii) Significant claustrophobia
8. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following injections or venepuncture.
9. Other major disease that, in the opinion of the Investigator, could interfere with a subject completing the study and necessary investigations.

2) Clinically significant smoking history. Defined as: Current smoker (any smoking including e-cigarettes in the last 3 months) or > 2 pack year smoking history at any time (2 pack years is equivalent to 20 cigarettes daily for 2 years), or use of any nicotine containing products, on more than one occasion, within the last 3 months.

3) History or presence of alcohol addiction, or excessive use of alcohol (average weekly intake in excess of 28 units alcohol; one unit being a half glass of beer, a small glass of wine or a measure of spirits)

4) Clinically significant history of use of drugs of misuse, with evidence of a negative drugs of misuse urine test required at screening and quarantine admission

5) History of anaphylaxis or any allergy likely to be worsened by any component of the study agent or proposed treatment regime.

6) Clinically active rhinitis (including hay fever) or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at time of inclusion into the study and/or requiring regular nasal corticosteroids on at least weekly basis, within 30 days of admission to quarantine.

7) Any significant abnormality altering the anatomy of the nose or nasopharynx, clinically significant history of epistaxis (nose bleeds) or any nasal or sinus surgery within six months of inoculation

8) Clinical, radiological, or laboratory evidence of current active TB disease or latent TB infection

9) Previous VZV pneumonia

10) Positive HBsAg, HCV or HIV antibodies

11) Concurrent use of oral, inhaled or systemic steroid medication or use within the last 6 months (steroids used as a cream or ointment are permissible), or the use of other immunosuppressive agents concurrently or within the last 6 months.

12) Concurrent use of medication contraindicated for use with Paxlovid rescue therapy

13) Administration of immunoglobulins and/or any blood products within the three months preceding the planned study challenge date

14) Current use of any medication or other drug taken through the nasal or inhaled route including cocaine or other recreational drugs

15) Plans to receive a live vaccination 30 days prior to enrolment, or any vaccination (i.e. non-live, including a SARS-CoV-2 vaccine) 21 days prior to enrolment and/or plans to take any vaccination 30 days following enrolment

16) Current pregnancy or pregnancy within the last 6 months, lactation or intention to become pregnant during study period

17) Shares a household with someone with clinically significant immunodeficiency (due to underlying medical condition, medication or pregnancy); or who is extremely clinically vulnerable (previously shielding under Public Health England (now referred to as UK HSA) guidelines)

18) Concurrent participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period

19) Laboratory confirmed (PCR or lateral flow antigen test) SARS-Cov-2 infection, evidence of viral pneumonitis on chest radiograph or a high clinical suspicion of COVID-19 disease in the 3 months preceding enrolment.

20) Post COVID-19 symptoms that have not resolved by 1 month prior to enrolment

21) Previous hospitalisation with COVID-19 disease or related complications e.g. pulmonary fibrosis on chest x ray

22) Family history of 1st degree relative aged 50 years or less with sudden cardiac or unexplained death

23) Family history of severe COVID-19 disease or response to any other viral disease e.g. Guillain-Barré

24) Family history unavailable or in opinion of investigators not sufficient to assess criteria 22 and 23.

25) Clinically significant abnormality on screening chest radiograph

26) Clinically significant abnormality of lung function testing

27) Clinically significant structural heart disease detected on CMR or echocardiogram, such as abnormal ventricular systolic function, evidence of previous myocardial infarction, previous myocarditis (on CMR) or significant valvular heart disease (more than mild)

28) Any clinically significant abnormality of screening blood or urine tests

29) Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data

30) Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.

For Groups 3 & 4:

31) Previous positive test for SARS CoV-2 infection (PCR or lateral flow antigen test) or a high clinical suspicion of COVID-19 disease at any time.

32) Positive Anti-nucleocapsid IgG at screening, unless explainable by vaccination

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited adverse events | Day 84
  To assess safety and human clinical response to wild type SARS-CoV-2 intranasal challenge in both previously SARS- CoV-2 infected (unvaccinated or vaccinated) and uninfected vaccinated participants via occurrence of adverse events (solicited and unsolicited) collected in e-diaries
Occurrence of adverse events as determined by medical assessment | Day 365
  Collection of AE data at each visit time point after SARS-CoV-2 inoculation (Graded 0-3)
Selection of optimal dose(s) | Day 14 or until discharge criteria is met
  The SARS-CoV-2 dose required to induce upper respiratory tract infection in 50% (+/-10%) of previously SARS-CoV-2 infected healthy volunteers following intranasal challenge.
  Defined by laboratory identification of SARS-CoV-2 from nasal and pharyngeal swab, using qPCR and/or quantitative live viral detection at two consecutive 12- hourly time points starting 24 hours post-inoculation and up to discharge from quarantine. Optimal dose to be defined in previously SARS-CoV-2 infected (vaccinated or unvaccinated) and uninfected vaccinated healthy volunteers

SECONDARY OUTCOMES:
Determination of SARS-CoV-2 viral dynamics | Day 365
  Assess the SARS-CoV-2 viral dynamics in upper respiratory samples from previously infected (vaccinated or unvaccinated) or uninfected vaccinated individuals including: determination of the incubation period, peak viral load and the mean duration of infectious viral shedding from quantitative virology measured using qPCR and/or live viral detection on naso-oropharyngeal samples.
Exploratory Immunology: Identification of laboratory markers | Day 365
  Ex-vivo ELISpot to SARS-CoV-2 peptide (sfc/1x10^6 PBMC)
Exploratory Immunology: Identification of laboratory markers | Day 365
  Innate, B cell and T cell flow cytometry panel to characterise surface cell markers and antigen specific responses to SARS-CoV-2 peptide before and after SARS-CoV-2 inoculation (% population)
Exploratory Immunology: Identification of laboratory markers | Day 365
  Neutralising peripheral blood antibody analysis to SARS-CoV-2
Exploratory Immunology: Identification of laboratory markers | Day 365
  Single cell RNA-seq on peripheral blood
Exploratory Immunology: Identification of laboratory markers | Day 365
  Cytokine analysis on serum and nasal mucosal lining fluid
Exploratory Immunology: Identification of laboratory markers | Day 365
  ELISA to SARS-CoV-2 peptide from serum and nasal mucosal lining fluid

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, MD and PhD, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Oxford Clinical Research Facility (OxCRF), Oxford, Oxon
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxon
  - Oxford University Hospital NHS Trust, Oxford, Oxon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson S, Marshall JL, Mawer A, Lopez-Ramon R, Harris SA, Satti I, Hughes E, Preston-Jones H, Cabrera Puig I, Longet S, Tipton T, Laidlaw S, Doherty RP, Morrison H, Mitchell R, Tanner R, Ateere A, Stylianou E, Wu MS, Fredsgaard-Jones TPW, Breuer J, Rapeport G, Ferreira VM, Gleeson F, Pollard AJ, Carroll M, Catchpole A, Chiu C, McShane H; COV-CHIM01 study team. Safety, tolerability, viral kinetics, and immune correlates of protection in healthy, seropositive UK adults inoculated with SARS-CoV-2: a single-centre, open-label, phase 1 controlled human infection study. Lancet Microbe. 2024 Jul;5(7):655-668. doi: 10.1016/S2666-5247(24)00025-9. Epub 2024 May 1. PMID 38703782